CLINICAL TRIAL: NCT01542138
Title: A Double Blind, Randomized Clinical Trial of 4% Niacinamide Versus 0.05% Desonide for the Treatment of Axillar Hyperpigmentation
Brief Title: Clinical Trial of 4% Niacinamide Versus 0.05% Desonide for the Treatment of Axillar Hyperpigmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Juan Pablo Castanedo Cazares, Dermatology research director, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIADESAH
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Hyperpigmentation
Keywords: Inflammatory hyperpigmentation, axillar pigmentation
MeSH Terms: conditions — Hyperpigmentation | interventions — Desonide; Niacinamide; nicomide; cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Niacinamide (Active Comparator): 4% niacinamide cream that will be randomly applied on axillar hyperpigmentation once-a-day for 9 weeks.
  Interventions: Drug: Niacinamide
- Desonide (Active Comparator): Once-a-day application of 0.05% desonide cream on axillar hyperpigmentation
  Interventions: Drug: Desonide
- Placebo (Placebo Comparator): Humectant placebo cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desonide — Once-a-day applying on axillar hyperpigmentation for 9 weeks
  Other Names: 0.05% Desowen cream, Galderma, France.
  Arms: Desonide
Drug: Niacinamide — Once-a-day applying on axillar hyperpigmentation for 9 weeks
  Other Names: Nicotinamide, nicomide
  Arms: Niacinamide
Drug: Placebo — Humectant placebo cream
  Other Names: vanicream, cetaphil
  Arms: Placebo

SUMMARY:
Axillary hyperpigmentation is a frequent consultation in dark skin populations although its exact prevalency is unknown. Currently, there are not studies about physiopathology and treatment for this entity. The objective is to evaluate the depigmenting effect of topical 4% niacinamide versus 0.05% desonide in axillary hyperpigmentation.

At least 30 axillas with hyperpigmentation in individuals of phototype III-V, aged 18-50 years are going to be randomly assigned to receive niacinamide, desonide or placebo daily. No hygienic habits will not be modified. Volunteers will be evaluated at baseline and for 9 weeks, by means of histological, histochemical and immunohistochemistry analysis, as well as Transepidermal Water Loss (TEWL), colorimetry, clinically and by photography control.

DETAILED DESCRIPTION:
Axillary hyperpigmentation is frequent in dark skin population, is possible a type of postinflammatory hyperpigmentation present in phototypes IV to VI. Previous reports have described increased intensity of Masson-Fontana, anti-tyrosinase and/or anti-TRP1 staining, indicative of melanocyte stimulation and increased melanin production, but the exact mechanism is unknown. The hair plucking, the rubbing of clothes on skin and physical stimulation from washing and drying the underarm are factors implicated. The objective of our study is evaluate the depigmenting effect of topical niacinamide versus desonide in axillary hyperpigmentation through the histochemistry and immunohistochemistry staining.

The study population will include at least 30 axillas with hyperpigmentation in a population with phototype III-V and aged 18-50 years old. Informed consent will be obtained from the patients, under approval by the local ethical committee (Institutional Review Board). The patients are going to be randomly assigned to receive 4% niacinamide, 0.05% desonide or placebo daily once at night. None hygienic habit is going to be modified. Volunteers will be evaluated at baseline and 9 weeks later, with histochemical and immunohistochemical analysis (biopsies), colorimetric value axis L*, a*, b* (Chromameter CR-300, Minolta, Osaka, Japan), Transepidermal Water Loss (TEWL) by means of an evaporimeter (Dermalab, Cortex Technology, Denmark), clinical assessment and photography control.

Statistical analysis was performed using t student, the level of significance was set at 5%. And clinical evaluation will be analysed by means of chi square test.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* Healthy
* Clinical diagnosis of axillar hyperpigmentation

Exclusion Criteria:

* Pregnancy or lactation
* Obesity
* Endocrinological diseases
* Mental diseases
* Treatment for axillar hyperpigmentation in the last 2 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pigmentation | 9 weeks
  Quantification of melanin content in histologic sections by Fontana-Masson stain

SECONDARY OUTCOMES:
Inflammation | 9 weeks
  Quantification of inflammatory infiltrate in skin biopsies by histologic lymphocites infiltrate and immunohistochemistry stain anti-CD1
Trauma | 9 weeks
  To detect trauma we measure damage in Membrane Basal by anti-collagen IV immunohistochemistry stain
Change in transepidermal water loss in hyperpigmented lesion | 9 weeks
  Quantification of water loss measured by a evaporimeter in grams per squared meter per hour. Is an indirect measure of inflammation.
Investigator's Depigmentation Improvement | 9 weeks
  Clinical improvement is assessed by means of digital photographic registration (frontal, right, and left views). Two independent observers clinically graded the global improvement as poor (0-25%), mild (26-50%), good (51-75%), and excellent (>75%).

CONTACTS AND LOCATIONS:
Overall Officials: Bertha Torres-Alvarez, MD, Study Chair — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosi, México; Gabryela N Larraga-Piñones, MD, Principal Investigator — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto". San Luis Potosi, México; Juan P Castanedo-Cázares, MD, Study Director — Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto". San Luis Potosi, México
Locations (1):
- Dermatology Department. Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Navarrete-Solis J, Castanedo-Cazares JP, Torres-Alvarez B, Oros-Ovalle C, Fuentes-Ahumada C, Gonzalez FJ, Martinez-Ramirez JD, Moncada B. A Double-Blind, Randomized Clinical Trial of Niacinamide 4% versus Hydroquinone 4% in the Treatment of Melasma. Dermatol Res Pract. 2011;2011:379173. doi: 10.1155/2011/379173. Epub 2011 Jul 21. PMID 21822427
- [Background] Torres-Alvarez B, Mesa-Garza IG, Castanedo-Cazares JP, Fuentes-Ahumada C, Oros-Ovalle C, Navarrete-Solis J, Moncada B. Histochemical and immunohistochemical study in melasma: evidence of damage in the basal membrane. Am J Dermatopathol. 2011 May;33(3):291-5. doi: 10.1097/DAD.0b013e3181ef2d45. PMID 21317614